CLINICAL TRIAL: NCT00306995
Title: A Phase III, Open, Randomized, Multicenter, Comparative Vaccination Study to Evaluate the Immunogenicity and Reactogenicity of Various Formulations of a Monovalent Candidate Pandemic Influenza A Vaccine in Individuals Over 60 Years of Age
Brief Title: Safety Study of Pandemic Candidate Influenza Vaccines in the Elderly Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102499
Record Dates: First submitted 2006-02-16; First posted 2006-03-27 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Influenza; Influenza Vaccines
Keywords: prophylaxis of pandemic influenza
MeSH Terms: conditions — Influenza, Human

ARMS (7):
- SB218352_15 Group (Experimental): Male and female subjects over 60 years of age, healthy or with underlying disease, received 2 doses of SB218352 pandemic influenza A formulation 1 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0 and Day 21.
  Interventions: Biological: SB218352_15
- SB218352_8 Group (Experimental): Male and female subjects over 60 years of age, healthy or with underlying disease, received 2 doses of SB218352 pandemic influenza A formulation 2 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0 and Day 21.
  Interventions: Biological: SB218352_8
- SB218352_4 Group (Experimental): Male and female subjects over 60 years of age, healthy or with underlying disease, received 2 doses of SB218352 pandemic influenza A formulation 3 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0 and Day 21.
  Interventions: Biological: SB218352_4
- SB218352_2 Group (Experimental): Male and female subjects over 60 years of age, healthy or with underlying disease, received 2 doses of SB218352 pandemic influenza A formulation 4 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0 and Day 21.
  Interventions: Biological: SB218352_2
- SB218352_8AL Group (Experimental): Male and female subjects over 60 years of age, healthy or with underlying disease, received 2 doses of SB218352 pandemic influenza A formulation 2 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0 and Day 21.
  Interventions: Biological: SB218352_8AL
- SB218352_4AL Group (Experimental): Male and female subjects over 60 years of age, healthy or with underlying disease, received 2 doses of SB218352 pandemic influenza A formulation 3 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0 and Day 21.
  Interventions: Biological: SB218352_4AL
- SB218352_2AL Group (Experimental): Male and female subjects over 60 years of age, healthy or with underlying disease, received 2 doses of SB218352 pandemic influenza A formulation 4 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0 and Day 21.
  Interventions: Biological: SB218352_2AL

INTERVENTIONS:
Biological: SB218352_15 — Non-adjuvanted pandemic influenza A formulation 1 vaccine
  Arms: SB218352_15 Group
Biological: SB218352_8 — Non-adjuvanted pandemic influenza A formulation 2 vaccine
  Arms: SB218352_8 Group
Biological: SB218352_4 — Non-adjuvanted pandemic influenza A formulation 3 vaccine
  Arms: SB218352_4 Group
Biological: SB218352_2 — Non-adjuvanted pandemic influenza A formulation 4 vaccine
  Arms: SB218352_2 Group
Biological: SB218352_8AL — Pandemic influenza A formulation 2 aluminium-adjuvanted vaccine
  Arms: SB218352_8AL Group
Biological: SB218352_4AL — Pandemic influenza A formulation 3 aluminium-adjuvanted vaccine
  Arms: SB218352_4AL Group
Biological: SB218352_2AL — Pandemic influenza A formulation 4 aluminium-adjuvanted vaccine
  Arms: SB218352_2AL Group

SUMMARY:
Influenza pandemics are caused by viruses that possess an Hemagglutinin molecule to which most of the population lacks immunity. If such virus is pathogenic to human and demonstrates the ability to transmit from person to person, the result is a global outbreak of disease that affects a high percentage of individuals in a short period of time and is likely to cause substantially increased mortality and morbidity in all countries of the world. Recently, purely avian influenza viruses, including the H5N1, H9N2 and H7N7 subtypes, have been directly transmitted to humans, raising concern over the possibility of a new influenza pandemic among the world's immunologically naive populations. In order to face this kind of situation, a pandemic influenza vaccine has to be developed.

ELIGIBILITY:
Inclusion criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol
* A male or female aged over 60 years at the time of vaccination.
* Written informed consent obtained from the subject.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Participation in an earlier study with a candidate pandemic H9N2 vaccine.
* Acute disease at the time of enrolment.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Drug and/or alcohol dependency.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2005-05-11 (Actual); Primary Completion 2006-07-04 (Actual); Study Completion 2006-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Germany (9):
  - GSK Investigational Site, Finsterwalde, Brandenburg
  - GSK Investigational Site, Ketzin, Brandenburg
  - GSK Investigational Site, Tostedt, Lower Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Geringswalde, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Elmshorn, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 102499 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102499 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102499 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102499 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102499 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After Part I, the core study (study period from Visit 1 on Day 0 up to the phone contact on Day 51), the enrolled subjects were stratified into Subset 1 (Part II - Visit 5 on Day 189 to study conclusion, i.e ., Visit 7 on Day 365) or Subset 2 (Part II - Visit 6 on Day 365 to study conclusion, i.e ., phone contact on Day 395).
Groups:
- SB218352_15 Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 1 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_8 Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_4 Group:: Male and fem le subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_2 Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_8AL Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at D y 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_4AL Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_2AL Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Da y 189 for subjects in Subs t I and at Day 0, Day 21 and Da y 365 for subjects in Subset 2.
Period: Study Part I
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Started | 55 | 55 | 55 | 55 | 55 | 55 | 55
Completed | 55 | 55 | 55 | 55 | 55 | 55 | 54
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Study Part II for Subset 1
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Started | 27 | 26 | 27 | 27 | 27 | 26 | 23
Completed | 27 | 26 | 27 | 27 | 27 | 26 | 23
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Study Part II for Subset 2
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Started | 23 | 24 | 23 | 22 | 23 | 26 | 24
Completed | 23 | 23 | 23 | 22 | 23 | 26 | 24
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Serious Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group: | Total
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55 | 55 | 385
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (5.11) | 69.0 (5.66) | 69.2 (5.77) | 69.1 (5.94) | 68.4 (5.92) | 68.4 (6.31) | 69.8 (5.91) | 68.9 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 30 | 32 | 28 | 41 | 22 | 212
  Male | 27 | 24 | 25 | 23 | 27 | 14 | 33 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Arabic/North African | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White-Caucasian | 55 | 55 | 55 | 54 | 55 | 55 | 55 | 384

OUTCOME MEASURES:

1. Primary Outcome: Serum Haemagglutination-inhibition (HI) Antibody Titers Against the Influenza A Virus Strain Subtype H9N2 (Anti-H9N2)
Description: Anti-H9N2 antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 10 post Dose 1
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- SB218352_2AL Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Titer | 24.4 [17.1 to 35.0] | 15.6 [11.0 to 22.1] | 14.6 [10.2 to 20.8] | 9.8 [7.5 to 12.8] | 23.3 [16.9 to 32.0] | 18.8 [12.3 to 28.5] | 16.9 [12.3 to 23.3]

2. Primary Outcome: Serum HI Antibody Titers Against the Influenza A Virus Strain Subtype H9N2 (Anti-H9N2)
Description: Anti-H9N2 antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 21 post Dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Titers | 32.5 [22.1 to 47.8] | 20.1 [14.0 to 28.9] | 21.9 [13.8 to 34.8] | 12.0 [9.1 to 15.9] | 42.1 [28.7 to 61.7] | 20.0 [13.3 to 30.0] | 17.8 [12.9 to 24.6]

3. Primary Outcome: Number of Seroconverted Subjects Against Influenza A Subtype H9N2
Description: Seroconversion rate was defined as the percentage of vaccinees who had a pre-vaccination HI titer lower than (<) 1:10 and a post-vaccination titre higher than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and a minimum four-fold increase in post-vaccination titer
Time Frame: At Day 10 post Dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Participants | 12 | 11 | 11 | 1 | 14 | 10 | 8

4. Primary Outcome: Number of Seroconverted Subjects Against Influenza A Subtype H9N2
Description: Seroconversion rate was defined as the percentage of vaccinees who had a pre-vaccination HI titer < 1:10 and a post-vaccination titre ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and a minimum four-fold increase in post-vaccination titer
Time Frame: At Day 21 post Dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Participants | 19 | 17 | 13 | 3 | 20 | 10 | 10

5. Primary Outcome: Seroconversion Factor for Influenza A Subtype H9N2
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs on day 10 compared to day 0.
Time Frame: At Day 10 post Dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Fold change | 2.7 [1.9 to 4.0] | 2.1 [1.5 to 3.0] | 2.0 [1.4 to 2.9] | 1.4 [1.2 to 1.7] | 3.1 [2.3 to 4.2] | 2.4 [1.6 to 3.7] | 2.4 [1.7 to 3.3]

6. Primary Outcome: Seroconversion Factor for Influenza A Subtype H9N2
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs on day 21 compared to day 0.
Time Frame: At Day 21 post Dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Fold change | 3.6 [2.3 to 5.7] | 2.7 [1.8 to 4.0] | 3.0 [1.8 to 5.0] | 1.7 [1.4 to 2.2] | 5.5 [3.7 to 8.4] | 2.6 [1.7 to 3.9] | 2.5 [1.8 to 3.5]

7. Primary Outcome: Number of Seroprotected Subjects Against H9N2
Description: Seroprotection rate was defined as the percentage of vaccinees with a serum HI titer ≥ 1:40 after vaccination (for each vaccine strain) that usually was accepted as indicating protection.
Time Frame: At Day 10 post Dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Participants | 19 | 13 | 14 | 6 | 20 | 16 | 11

8. Primary Outcome: Number of Seroprotected Subjects Against H9N2
Description: as for outcome 7
Time Frame: At Day 21 post Dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Participants | 24 | 19 | 16 | 7 | 27 | 15 | 13

9. Primary Outcome: Number of Subjects With Seroprotection Power Against H9N2
Description: Seroprotection power was defined as the proportion of subjects who were unprotected prior to the vaccination (HI titer < 1:40 on day 0) and had a protective post-vaccination titer of ≥ 1:40.
Time Frame: At Day 10 post Dose 1
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence, which included all evaluable subjects for whom data concerning persistence of the immune response induced by the vaccine were available for the specified time points.
Measure: Count of Participants; unit: Participants
Groups:
- SB218352_15 Subset 1: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 1 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189.
- SB218352_8 Subset 1: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189.
- SB218352_4 Subset 1: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189.
- SB218352_2 Subset 1: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189.
- SB218352_8AL Subset 1: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189.
- SB218352_4AL Subset 1: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189.
- SB218352_2AL Subset 1: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189.
- SB218352_15 Subset 2: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 1 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 365.
- SB218352_8 Subset 2: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 365.
- SB218352_4 Subset 2: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 365.
- SB218352_2 Subset 2: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 365.
- SB218352_8AL Subset 2: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 365.
- SB218352_4AL Subset 2: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 365.
- SB218352_2AL Subset 2: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 365.
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 22 | 25 | 26 | 25 | 25 | 25 | 23 | 21 | 22 | 20 | 18 | 20 | 24 | 21
Participants | 4 | 4 | 6 | 2 | 5 | 7 | 0 | 8 | 7 | 4 | 0 | 10 | 7 | 7

10. Primary Outcome: Number of Subjects With Seroprotection Power Against H9N2
Description: as for outcome 9
Time Frame: At Day 21 post Dose 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 22 | 25 | 26 | 25 | 25 | 25 | 22 | 21 | 22 | 20 | 18 | 20 | 24 | 21
Participants | 7 | 9 | 8 | 3 | 8 | 7 | 1 | 9 | 8 | 4 | 0 | 12 | 6 | 8

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-days (Day 0-30) post vaccination
Population: The analysis was performed on the Total Vaccinated Cohort (TVc), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- SB218352_4 Group:: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55 | 55
Participants
  Any AEs | 8 | 3 | 3 | 6 | 4 | 4 | 7
  Grade 3 AEs | 2 | 0 | 1 | 0 | 0 | 0 | 1
  Related AEs | 1 | 1 | 0 | 0 | 0 | 1 | 2

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: A SAE was any untoward medical occurrence which resulted in death, was life-threatening, resulted in hospitalization or prolongation of hospitalization, resulted in permanent of serious physical disability or incapacity, caused a congenital anomaly or birth defect in the offspring of a subject or might have put the subject at risk based on medical or scientific judgment or necessitated intervention to prevent such an event (e.q. invasive or malignant cancers, intensive treatment in an emergency room or at home for bronchospasm, blood dyscrasias, or convulsion that do not resulted in hospitalization).
Time Frame: From Day 0 to Day 51
Population: The analysis was performed on the Total Vaccinated Cohort (TVc), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55 | 55
Participants | 1 | 0 | 1 | 0 | 0 | 0 | 1

13. Secondary Outcome: Frequency of Antigen-specific Cluster of Differentiation 4 (CD4) T-cells
Description: Among expressed immune markers were interferon-gamma (IFN-γ) and cluster of differentiation 40 - ligand (CD40-L).
Time Frame: At Days 0, 10, 21 and 42 post vaccination
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 23 | 25 | 23 | 26 | 27 | 22 | 24
T-cells/million cells
  CD4-ALL DOUBLES, Day 0: number analyzed (Participants) | 23 | 25 | 23 | 25 | 27 | 22 | 24
  CD4-ALL DOUBLES, Day 0 | 557.00 [509.00 to 827.00] | 785.00 [489.00 to 1072.00] | 782.00 [441.00 to 1052.00] | 472.00 [305.00 to 1025.00] | 738.00 [558.00 to 1284.00] | 691.00 [547.00 to 873.00] | 594.50 [453.50 to 1020.50]
  CD4-ALL DOUBLES, DAY 10: number analyzed (Participants) | 23 | 21 | 22 | 23 | 25 | 21 | 21
  CD4-ALL DOUBLES, DAY 10 | 1049.00 [779.00 to 1753.00] | 1148.00 [702.00 to 1891.00] | 1066.50 [647.00 to 1809.00] | 844.00 [478.00 to 1548.00] | 1275.00 [884.00 to 1691.00] | 1194.00 [760.00 to 1453.00] | 874.00 [626.00 to 1399.00]
  CD4-ALL DOUBLES, DAY 21: number analyzed (Participants) | 23 | 22 | 21 | 26 | 23 | 20 | 22
  CD4-ALL DOUBLES, DAY 21 | 1118.00 [904.00 to 1424.00] | 1396.00 [923.00 to 1962.00] | 1212.00 [784.00 to 1822.00] | 791.50 [390.00 to 1229.00] | 1555.00 [1073.00 to 1873.00] | 989.50 [734.00 to 1912.50] | 972.50 [820.00 to 1466.00]
  CD4-ALL DOUBLES, DAY 42: number analyzed (Participants) | 21 | 23 | 19 | 23 | 24 | 20 | 22
  CD4-ALL DOUBLES, DAY 42 | 1100.00 [733.00 to 1567.00] | 1349.00 [722.00 to 1812.00] | 967.00 [647.00 to 1693.00] | 965.00 [651.00 to 1645.00] | 1600.00 [936.00 to 2156.00] | 1198.00 [791.50 to 1646.50] | 1059.50 [894.00 to 1636.00]
  CD4-CD40L, Day 0: number analyzed (Participants) | 23 | 25 | 23 | 25 | 27 | 22 | 24
  CD4-CD40L, Day 0 | 583.00 [471.00 to 810.00] | 574.00 [467.00 to 1095.00] | 750.00 [441.00 to 1028.00] | 438.00 [308.00 to 920.00] | 720.00 [442.00 to 1263.00] | 714.00 [368.00 to 866.00] | 600.00 [449.00 to 976.00]
  CD4-CD40L, DAY 10: number analyzed (Participants) | 23 | 21 | 22 | 23 | 25 | 21 | 21
  CD4-CD40L, DAY 10 | 1028.00 [779.00 to 1446.00] | 1148.00 [668.00 to 1922.00] | 981.00 [626.00 to 1654.00] | 769.00 [478.00 to 1552.00] | 1161.00 [630.00 to 1639.00] | 1158.00 [760.00 to 1378.00] | 886.00 [613.00 to 1399.00]
  CD4-CD40L, DAY 21: number analyzed (Participants) | 23 | 22 | 21 | 26 | 23 | 20 | 22
  CD4-CD40L, DAY 21 | 1069.00 [851.00 to 1320.00] | 1243.50 [730.00 to 1511.00] | 1074.00 [752.00 to 1483.00] | 788.50 [376.00 to 1229.00] | 1536.00 [884.00 to 1820.00] | 974.50 [710.00 to 1790.00] | 900.50 [753.00 to 1421.00]
  CD4-CD40L, DAY 42: number analyzed (Participants) | 21 | 23 | 19 | 23 | 24 | 20 | 22
  CD4-CD40L, DAY 42 | 1037.00 [721.00 to 1545.00] | 1088.00 [649.00 to 1748.00] | 945.00 [641.00 to 1644.00] | 999.00 [651.00 to 1645.00] | 1492.50 [836.00 to 2147.50] | 1177.50 [746.50 to 1608.50] | 984.00 [824.00 to 1636.00]
  CD4-IFN-γ, Day 0: number analyzed (Participants) | 23 | 25 | 23 | 25 | 27 | 22 | 24
  CD4-IFN-γ, Day 0 | 278.00 [120.00 to 353.00] | 233.00 [109.00 to 761.00] | 198.00 [172.00 to 395.00] | 160.00 [80.00 to 280.00] | 299.00 [125.00 to 434.00] | 212.50 [177.00 to 464.00] | 217.50 [149.00 to 295.50]
  CD4-IFN-γ, DAY 10: number analyzed (Participants) | 23 | 21 | 22 | 23 | 25 | 21 | 21
  CD4-IFN-γ, DAY 10 | 466.00 [273.00 to 612.00] | 457.00 [196.00 to 539.00] | 582.50 [336.00 to 693.00] | 365.00 [93.00 to 674.00] | 463.00 [239.00 to 926.00] | 400.00 [170.00 to 581.00] | 245.00 [196.00 to 425.00]
  CD4-IFN-γ, DAY 21: number analyzed (Participants) | 23 | 22 | 21 | 26 | 23 | 20 | 22
  CD4-IFN-γ, DAY 21 | 411.00 [231.00 to 638.00] | 482.00 [253.00 to 651.00] | 516.00 [291.00 to 629.00] | 228.50 [171.00 to 558.00] | 484.00 [305.00 to 784.00] | 391.00 [204.00 to 911.50] | 412.00 [298.00 to 654.00]
  CD4-IFN-γ, DAY 42: number analyzed (Participants) | 21 | 23 | 19 | 23 | 24 | 20 | 22
  CD4-IFN-γ, DAY 42 | 342.00 [234.00 to 449.00] | 332.00 [245.00 to 739.00] | 346.00 [232.00 to 549.00] | 344.00 [211.00 to 632.00] | 669.50 [312.50 to 915.50] | 445.00 [361.50 to 790.00] | 483.00 [232.00 to 733.00]

14. Secondary Outcome: Frequency of Antigen-specific CD4 T-cells
Description: Among expressed immune markers were interleukin-2 (IL-2) and tumour necrosis factor-alpha (TNF-α).
Time Frame: At Days 0, 10, 21 and 42 post-vaccination
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 23 | 25 | 23 | 26 | 27 | 22 | 24
T-cells/million cells
  CD4-IL-2, DAY 0: number analyzed (Participants) | 23 | 25 | 23 | 25 | 27 | 22 | 24
  CD4-IL-2, DAY 0 | 414.00 [322.00 to 661.00] | 491.00 [356.00 to 922.00] | 524.00 [351.00 to 801.00] | 381.00 [208.00 to 559.00] | 509.00 [377.00 to 987.00] | 487.50 [269.00 to 579.00] | 437.00 [320.00 to 641.50]
  CD4-IL-2, DAY 10: number analyzed (Participants) | 23 | 21 | 22 | 23 | 25 | 21 | 21
  CD4-IL-2, DAY 10 | 751.00 [582.00 to 1234.00] | 985.00 [581.00 to 1423.00] | 814.00 [460.00 to 1271.00] | 579.00 [264.00 to 1106.00] | 924.00 [619.00 to 1284.00] | 821.00 [616.00 to 1155.00] | 622.00 [392.00 to 981.00]
  CD4-IL-2, DAY 21: number analyzed (Participants) | 23 | 22 | 21 | 26 | 23 | 20 | 22
  CD4-IL-2, DAY 21 | 888.00 [557.00 to 1221.00] | 1013.50 [819.00 to 1790.00] | 814.00 [569.00 to 1281.00] | 625.00 [227.00 to 865.00] | 988.00 [763.00 to 1697.00] | 799.00 [640.00 to 1405.50] | 764.00 [632.00 to 1070.00]
  CD4-IL-2, DAY 42: number analyzed (Participants) | 21 | 23 | 19 | 23 | 24 | 20 | 22
  CD4-IL-2, DAY 42 | 913.00 [561.00 to 1334.00] | 876.00 [562.00 to 1529.00] | 714.00 [559.00 to 1322.00] | 761.00 [534.00 to 1224.00] | 1233.50 [707.50 to 1743.50] | 953.00 [658.50 to 1331.00] | 890.00 [583.00 to 1216.00]
  CD4-TNF-α, DAY 0: number analyzed (Participants) | 23 | 25 | 23 | 25 | 27 | 22 | 24
  CD4-TNF-α, DAY 0 | 380.00 [273.00 to 669.00] | 470.00 [287.00 to 999.00] | 495.00 [321.00 to 676.00] | 337.00 [240.00 to 705.00] | 538.00 [327.00 to 759.00] | 495.50 [348.00 to 669.00] | 395.00 [282.00 to 680.50]
  CD4-TNF-α, DAY 10: number analyzed (Participants) | 23 | 21 | 22 | 23 | 25 | 21 | 21
  CD4-TNF-α, DAY 10 | 817.00 [665.00 to 1229.00] | 822.00 [491.00 to 1141.00] | 717.00 [347.00 to 1062.00] | 522.00 [376.00 to 1073.00] | 728.00 [534.00 to 1126.00] | 793.00 [637.00 to 875.00] | 641.00 [414.00 to 929.00]
  CD4-TNF-α, DAY 21: number analyzed (Participants) | 23 | 22 | 21 | 26 | 23 | 20 | 22
  CD4-TNF-α, DAY 21 | 923.00 [637.00 to 1207.00] | 842.50 [676.00 to 1303.00] | 870.00 [519.00 to 1252.00] | 491.50 [359.00 to 837.00] | 1244.00 [749.00 to 1455.00] | 650.50 [458.50 to 1307.50] | 672.50 [557.00 to 1150.00]
  CD4-TNF-α, DAY 42: number analyzed (Participants) | 21 | 23 | 19 | 23 | 24 | 20 | 22
  CD4-TNF-α, DAY 42 | 868.00 [530.00 to 1163.00] | 899.00 [505.00 to 1436.00] | 608.00 [464.00 to 994.00] | 717.00 [368.00 to 1261.00] | 1079.50 [696.50 to 1621.00] | 829.00 [592.50 to 1128.50] | 722.00 [520.00 to 988.00]

15. Secondary Outcome: Cytokine-positive CD4 T-cells Frequency
Description: Among expressed immune markers were interleukin-2 (IL-2), interferon-gamma (IFN-γ), tumour necrosis factor-alpha (TNF-α) and cluster of differentiation 40 - ligand (CD40-L). Descriptive comparison of the CMI response after Dose 1 and Dose 2 of the monovalent candidate pandemic influenza A vaccine. CMI response was determined in terms of the proportion of lymphocytes (CD4+ and CD8+ per million T cells) activated in vitro by the vaccine antigen on Days 10 and 21 after the Dose 1 and on Day 21 after Dose 2 as compared to Day 0 (pre-vaccination). The results were calculated based on the individual difference between each post-vaccination timepoint (Day 10, Day 21, Day 42) and Day 0.
Time Frame: At Days 10, 21 and 42 post-vaccination
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 21 | 21 | 20 | 24 | 24 | 19 | 21
CD4+ T-cells/million cells
  CD4-ALL DOUBLES, DAY 10: number analyzed (Participants) | 21 | 20 | 20 | 22 | 24 | 19 | 20
  CD4-ALL DOUBLES, DAY 10 | 295.00 [9.00 to 859.00] | 326.00 [127.50 to 731.00] | 219.00 [-64.00 to 767.00] | 342.00 [-58.00 to 657.00] | 434.50 [24.00 to 796.50] | 398.00 [11.00 to 773.00] | 139.00 [-69.50 to 981.00]
  CD4-ALL DOUBLES, DAY 21: number analyzed (Participants) | 21 | 20 | 19 | 24 | 22 | 18 | 21
  CD4-ALL DOUBLES, DAY 21 | 248.00 [108.00 to 539.00] | 477.00 [280.50 to 766.00] | 359.00 [-114.00 to 780.00] | 252.50 [-62.00 to 669.00] | 645.00 [274.00 to 1037.00] | 440.50 [177.00 to 1195.00] | 283.00 [98.00 to 660.00]
  CD4-ALL DOUBLES, DAY 42: number analyzed (Participants) | 18 | 21 | 16 | 21 | 23 | 17 | 20
  CD4-ALL DOUBLES, DAY 42 | 384.00 [116.00 to 678.00] | 360.00 [-120.00 to 766.00] | 482.50 [-3.00 to 791.00] | 441.00 [298.00 to 708.00] | 689.00 [9.00 to 1104.00] | 554.00 [353.00 to 751.00] | 445.50 [252.50 to 786.50]
  CD4-CD40L, DAY 10: number analyzed (Participants) | 21 | 20 | 20 | 22 | 24 | 19 | 20
  CD4-CD40L, DAY 10 | 302.00 [-18.00 to 859.00] | 299.50 [20.50 to 680.50] | 149.50 [-98.50 to 686.50] | 303.50 [-28.00 to 650.00] | 384.50 [10.50 to 745.50] | 335.00 [-9.00 to 741.00] | 104.50 [-37.00 to 930.00]
  CD4-CD40L, DAY 21: number analyzed (Participants) | 21 | 20 | 19 | 24 | 22 | 18 | 21
  CD4-CD40L, DAY 21 | 195.00 [4.00 to 481.00] | 429.50 [142.00 to 623.00] | 271.00 [-114.00 to 735.00] | 237.00 [-42.50 to 639.50] | 630.00 [48.00 to 996.00] | 433.00 [158.00 to 1095.00] | 286.00 [70.00 to 547.00]
  CD4-CD40L, DAY 42: number analyzed (Participants) | 18 | 21 | 16 | 21 | 23 | 17 | 20
  CD4-CD40L, DAY 42 | 228.00 [62.00 to 687.00] | 320.00 [-14.00 to 737.00] | 440.00 [-88.00 to 691.00] | 451.00 [310.00 to 751.00] | 685.00 [-3.00 to 1071.00] | 513.00 [336.00 to 725.00] | 445.00 [232.50 to 765.00]
  CD4-IFN-γ, DAY 10: number analyzed (Participants) | 21 | 20 | 20 | 22 | 24 | 19 | 20
  CD4-IFN-γ, DAY 10 | 105.00 [-17.00 to 200.00] | 134.50 [-108.00 to 451.50] | 172.50 [3.50 to 478.00] | 78.50 [0.00 to 438.00] | 167.00 [92.00 to 427.00] | 165.00 [23.00 to 273.00] | 72.50 [-54.50 to 375.00]
  CD4-IFN-γ, DAY 21: number analyzed (Participants) | 21 | 20 | 19 | 24 | 22 | 18 | 21
  CD4-IFN-γ, DAY 21 | 107.00 [-58.00 to 256.00] | 120.00 [-34.00 to 442.00] | 205.00 [-3.00 to 343.00] | 77.50 [-41.00 to 304.00] | 145.50 [57.00 to 506.00] | 229.00 [-57.00 to 600.00] | 150.00 [83.00 to 260.00]
  CD4-IFN-γ, DAY 42: number analyzed (Participants) | 18 | 21 | 16 | 21 | 23 | 17 | 20
  CD4-IFN-γ, DAY 42 | 125.00 [27.00 to 196.00] | 145.00 [-115.00 to 236.00] | 124.00 [8.50 to 350.50] | 136.00 [60.00 to 248.00] | 320.00 [-19.00 to 621.00] | 186.00 [103.00 to 375.00] | 233.50 [64.50 to 544.00]
  CD4-IL-2, DAY 10: number analyzed (Participants) | 21 | 20 | 20 | 22 | 24 | 19 | 20
  CD4-IL-2, DAY 10 | 226.00 [51.00 to 574.00] | 289.50 [48.00 to 729.50] | 152.00 [-45.50 to 648.50] | 225.00 [0.00 to 442.00] | 369.50 [-38.00 to 645.00] | 242.00 [120.00 to 668.00] | 158.50 [-90.00 to 523.00]
  CD4-IL2, DAY 21: number analyzed (Participants) | 21 | 20 | 19 | 24 | 22 | 18 | 21
  CD4-IL2, DAY 21 | 227.00 [48.00 to 547.00] | 401.00 [170.50 to 644.00] | 297.00 [15.00 to 549.00] | 117.00 [-64.50 to 459.00] | 400.50 [132.00 to 789.00] | 518.00 [224.00 to 701.00] | 257.00 [150.00 to 499.00]
  CD4-IL-2, DAY 42: number analyzed (Participants) | 18 | 21 | 16 | 21 | 23 | 17 | 20
  CD4-IL-2, DAY 42 | 363.50 [57.00 to 613.00] | 285.00 [58.00 to 540.00] | 294.50 [158.00 to 457.50] | 359.00 [180.00 to 656.00] | 648.00 [40.00 to 970.00] | 523.00 [381.00 to 629.00] | 493.00 [198.00 to 766.50]
  CD4-TNF-α, DAY 10: number analyzed (Participants) | 21 | 20 | 20 | 22 | 24 | 19 | 20
  CD4-TNF-α, DAY 10 | 324.00 [50.00 to 425.00] | 221.50 [41.00 to 608.50] | 194.00 [70.50 to 550.00] | 122.00 [-68.00 to 501.00] | 210.50 [-61.00 to 423.00] | 194.00 [-33.00 to 469.00] | 140.50 [-42.00 to 540.50]
  CD4-TNF-α, DAY 21: number analyzed (Participants) | 21 | 20 | 19 | 24 | 22 | 18 | 21
  CD4-TNF-α, DAY 21 | 293.00 [150.00 to 412.00] | 282.50 [164.00 to 610.50] | 259.00 [12.00 to 648.00] | 142.50 [-17.00 to 430.00] | 470.50 [233.00 to 795.00] | 156.50 [31.00 to 937.00] | 229.00 [139.00 to 340.00]
  CD4-TNF-α, DAY 42: number analyzed (Participants) | 18 | 21 | 16 | 21 | 23 | 17 | 20
  CD4-TNF-α, DAY 42 | 291.50 [177.00 to 693.00] | 157.00 [-46.00 to 538.00] | 175.00 [-20.50 to 510.50] | 239.00 [114.00 to 574.00] | 454.00 [234.00 to 805.00] | 313.00 [239.00 to 484.00] | 252.50 [106.00 to 606.00]

16. Secondary Outcome: Frequency of Antigen-specific Cluster of Differentiation 8 (CD8) T-cells
Description: Among expressed immune markers were interferon-gamma (IFN-γ) and cluster of differentiation 40 - ligand (CD40-L).
Time Frame: At Days 0, 10, 21 and 42 post-vaccination
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 26 | 22 | 22
CD8+ T-cells/million cells
  CD8-ALL DOUBLES, Day 0: number analyzed (Participants) | 21 | 24 | 23 | 22 | 26 | 22 | 22
  CD8-ALL DOUBLES, Day 0 | 107.00 [1.00 to 168.00] | 62.00 [1.00 to 186.00] | 104.00 [27.00 to 292.00] | 83.50 [1.00 to 294.00] | 83.00 [1.00 to 302.00] | 83.00 [1.00 to 263.00] | 12.00 [1.00 to 124.00]
  CD8-ALL DOUBLES, DAY 10: number analyzed (Participants) | 20 | 18 | 22 | 21 | 24 | 18 | 20
  CD8-ALL DOUBLES, DAY 10 | 104.50 [1.00 to 320.00] | 47.50 [1.00 to 195.00] | 148.00 [2.00 to 218.00] | 102.00 [1.00 to 235.00] | 34.00 [1.00 to 313.00] | 73.00 [9.00 to 347.00] | 17.50 [1.00 to 175.00]
  CD8-ALL DOUBLES, DAY 21: number analyzed (Participants) | 16 | 19 | 21 | 23 | 19 | 17 | 18
  CD8-ALL DOUBLES, DAY 21 | 76.00 [1.00 to 187.50] | 19.00 [1.00 to 151.00] | 57.00 [1.00 to 361.00] | 51.00 [1.00 to 378.00] | 172.00 [1.00 to 482.00] | 98.00 [1.00 to 304.00] | 1.00 [1.00 to 265.00]
  CD8-ALL DOUBLES, DAY 42: number analyzed (Participants) | 12 | 19 | 14 | 18 | 19 | 18 | 16
  CD8-ALL DOUBLES, DAY 42 | 17.50 [1.00 to 438.50] | 70.00 [1.00 to 258.00] | 167.50 [43.00 to 336.00] | 147.50 [1.00 to 301.00] | 163.00 [1.00 to 307.00] | 173.50 [1.00 to 434.00] | 100.00 [1.00 to 358.00]
  CD8-CD40L, Day 0: number analyzed (Participants) | 21 | 24 | 23 | 22 | 26 | 22 | 22
  CD8-CD40L, Day 0 | 1.00 [1.00 to 54.00] | 1.00 [1.00 to 58.50] | 49.00 [1.00 to 101.00] | 1.00 [1.00 to 52.00] | 1.00 [1.00 to 60.00] | 1.00 [1.00 to 102.00] | 1.00 [1.00 to 113.00]
  CD8-CD40L, DAY 10: number analyzed (Participants) | 20 | 18 | 22 | 21 | 24 | 18 | 20
  CD8-CD40L, DAY 10 | 1.50 [1.00 to 81.50] | 1.00 [1.00 to 4.00] | 3.50 [1.00 to 60.00] | 1.00 [1.00 to 190.00] | 1.00 [1.00 to 95.50] | 49.50 [1.00 to 98.00] | 1.00 [1.00 to 9.50]
  CD8-CD40L, DAY 21: number analyzed (Participants) | 16 | 19 | 21 | 23 | 19 | 17 | 18
  CD8-CD40L, DAY 21 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 52.00] | 51.00 [1.00 to 82.00] | 1.00 [1.00 to 7.00] | 1.00 [1.00 to 56.00] | 1.00 [1.00 to 51.00] | 1.00 [1.00 to 49.00]
  CD8-CD40L, DAY 42: number analyzed (Participants) | 12 | 19 | 14 | 18 | 19 | 18 | 16
  CD8-CD40L, DAY 42 | 1.00 [1.00 to 100.00] | 1.00 [1.00 to 49.00] | 48.00 [1.00 to 101.00] | 25.50 [1.00 to 97.00] | 1.00 [1.00 to 78.00] | 26.50 [1.00 to 135.00] | 3.50 [1.00 to 149.50]
  CD8-IFN-γ, Day 0: number analyzed (Participants) | 21 | 24 | 23 | 22 | 26 | 22 | 22
  CD8-IFN-γ, Day 0 | 1.00 [1.00 to 107.00] | 21.50 [1.00 to 108.00] | 97.00 [1.00 to 204.00] | 1.00 [1.00 to 103.00] | 52.50 [1.00 to 150.00] | 50.50 [1.00 to 155.00] | 1.00 [1.00 to 113.00]
  CD8-IFN-γ, DAY 10: number analyzed (Participants) | 20 | 18 | 22 | 21 | 24 | 18 | 20
  CD8-IFN-γ, DAY 10 | 68.00 [1.00 to 156.00] | 1.00 [1.00 to 50.00] | 1.00 [1.00 to 131.00] | 50.00 [1.00 to 155.00] | 49.50 [1.00 to 167.50] | 48.50 [1.00 to 141.00] | 49.00 [1.00 to 192.50]
  CD8-IFN-γ, DAY 21: number analyzed (Participants) | 16 | 19 | 21 | 23 | 19 | 17 | 18
  CD8-IFN-γ, DAY 21 | 15.50 [1.00 to 159.00] | 1.00 [1.00 to 76.00] | 54.00 [1.00 to 155.00] | 29.00 [1.00 to 107.00] | 50.00 [1.00 to 303.00] | 49.00 [1.00 to 128.00] | 1.00 [1.00 to 51.00]
  CD8-IFN-γ, DAY 42: number analyzed (Participants) | 12 | 19 | 14 | 18 | 19 | 18 | 16
  CD8-IFN-γ, DAY 42 | 25.00 [1.00 to 122.50] | 1.00 [1.00 to 130.00] | 60.00 [1.00 to 111.00] | 82.00 [1.00 to 277.00] | 98.00 [1.00 to 313.00] | 94.50 [1.00 to 129.00] | 50.50 [1.00 to 198.50]

17. Secondary Outcome: Frequency of Antigen-specific CD8 T-cells
Description: Among expressed immune markers were interleukin-2 (IL-2) and tumour necrosis factor-alpha (TNF-α).
Time Frame: At Days 0, 10, 21 and 42 post-vaccination
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Groups:
- SB218352_15 Group: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 1 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_8 Group: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_4 Group: Male and fem le subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm , at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_2 Group: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 non-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_8AL Group: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 2 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-dominant arm, at D y 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_4AL Group: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 3 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-domina nt arm, at Day 0, Day 21 and Day 189 for subjects in Subset I and at Day 0, Day 21 and Day 365 for subjects in Subset 2.
- SB218352_2AL Group: Male and female subjects over 60 years of age, healthy or with underlying disease, received 3 doses of SB218352 pandemic influenza A formulation 4 aluminium-adjuvanted vaccine, administered in the deltoid region of the non-domina nt arm, at Day 0, Day 21 and Da y 189 for subjects in Subs t I and at Day 0, Day 21 and Da y 365 for subjects in Subset 2.
Arm/Group | SB218352_15 Group | SB218352_8 Group | SB218352_4 Group | SB218352_2 Group | SB218352_8AL Group | SB218352_4AL Group | SB218352_2AL Group
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 26 | 22 | 22
CD8+ T-cells/million cells
  CD8-IL-2, Day 0: number analyzed (Participants) | 21 | 24 | 23 | 22 | 26 | 22 | 22
  CD8-IL-2, Day 0 | 52.00 [1.00 to 152.00] | 20.00 [1.00 to 128.00] | 56.00 [1.00 to 238.00] | 34.50 [1.00 to 198.00] | 7.50 [1.00 to 90.00] | 25.00 [1.00 to 179.00] | 4.00 [1.00 to 62.00]
  CD8-IL-2, DAY 10: number analyzed (Participants) | 20 | 18 | 22 | 21 | 24 | 18 | 20
  CD8-IL-2, DAY 10 | 27.50 [1.00 to 154.50] | 1.00 [1.00 to 195.00] | 50.00 [1.00 to 166.00] | 64.00 [1.00 to 235.00] | 1.50 [1.00 to 155.00] | 71.50 [1.00 to 231.00] | 1.00 [1.00 to 100.00]
  CD8-IL-2, DAY 21: number analyzed (Participants) | 16 | 19 | 21 | 23 | 19 | 17 | 18
  CD8-IL-2, DAY 21 | 1.00 [1.00 to 46.00] | 19.00 [1.00 to 97.00] | 1.00 [1.00 to 192.00] | 23.00 [1.00 to 211.00] | 24.00 [1.00 to 173.00] | 38.00 [1.00 to 304.00] | 1.00 [1.00 to 73.00]
  CD8-IL-2, DAY 42: number analyzed (Participants) | 12 | 19 | 14 | 18 | 19 | 18 | 16
  CD8-IL-2, DAY 42 | 49.50 [1.00 to 291.50] | 1.00 [1.00 to 260.00] | 98.50 [1.00 to 248.00] | 24.50 [1.00 to 151.00] | 47.00 [1.00 to 153.00] | 29.50 [1.00 to 365.00] | 25.00 [1.00 to 262.00]
  CD8-TNF-α, Day 0 | 60.00 [1.00 to 105.00] | 19.50 [1.00 to 154.50] | 51.00 [1.00 to 241.00] | 50.00 [1.00 to 155.00] | 85.50 [10.00 to 267.00] | 77.00 [1.00 to 155.00] | 10.50 [1.00 to 96.00]
  CD8-TNF-α, DAY 10: number analyzed (Participants) | 20 | 18 | 22 | 21 | 24 | 18 | 20
  CD8-TNF-α, DAY 10 | 107.50 [1.00 to 242.00] | 25.00 [1.00 to 150.00] | 77.00 [1.00 to 171.00] | 49.00 [1.00 to 198.00] | 82.00 [1.00 to 210.00] | 51.50 [1.00 to 198.00] | 1.00 [1.00 to 124.00]
  CD8-TNF-α, DAY 21: number analyzed (Participants) | 16 | 19 | 21 | 23 | 19 | 17 | 18
  CD8-TNF-α, DAY 21 | 75.00 [1.00 to 272.50] | 51.00 [1.00 to 100.00] | 57.00 [1.00 to 220.00] | 23.00 [1.00 to 374.00] | 100.00 [1.00 to 388.00] | 48.00 [1.00 to 289.00] | 1.00 [1.00 to 97.00]
  CD8-TNF-α, DAY 42: number analyzed (Participants) | 12 | 19 | 14 | 18 | 19 | 18 | 16
  CD8-TNF-α, DAY 42 | 29.50 [1.00 to 386.50] | 101.00 [1.00 to 258.00] | 157.00 [50.00 to 226.00] | 76.00 [1.00 to 301.00] | 163.00 [1.00 to 307.00] | 110.00 [3.00 to 434.00] | 49.00 [1.00 to 163.50]

18. Secondary Outcome: Cytokine-positive CD8 T-cells Frequency
Description: as for outcome 15
Time Frame: At Days 10, 21 and 42 post-vaccination
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | SB218352_15 Group | SB218352_8 Group | SB218352_4 Group | SB218352_2 Group | SB218352_8AL Group | SB218352_4AL Group | SB218352_2AL Group
Number analyzed (Participants) | 17 | 17 | 20 | 19 | 22 | 16 | 17
CD8+ T-cells/million cells
  CD8-ALL DOUBLES, DAY 10: number analyzed (Participants) | 17 | 17 | 20 | 18 | 22 | 16 | 17
  CD8-ALL DOUBLES, DAY 10 | 2.00 [-86.00 to 143.00] | 0.00 [-99.00 to 47.00] | 16.00 [-145.00 to 152.00] | 0.00 [-50.00 to 100.00] | 0.00 [-234.00 to 155.00] | 4.00 [-155.00 to 267.00] | 0.00 [-21.00 to 49.00]
  CD8-ALL DOUBLES, DAY 21: number analyzed (Participants) | 14 | 17 | 19 | 19 | 17 | 15 | 16
  CD8-ALL DOUBLES, DAY 21 | -46.00 [-118.00 to 85.00] | 0.00 [-126.00 to 51.00] | -31.00 [-266.00 to 105.00] | 0.00 [-45.00 to 223.00] | 0.00 [-98.00 to 1.00] | 0.00 [-48.00 to 218.00] | 0.00 [-37.00 to 59.50]
  CD8-ALL DOUBLES, DAY 42: number analyzed (Participants) | 10 | 17 | 11 | 15 | 17 | 15 | 14
  CD8-ALL DOUBLES, DAY 42 | -50.50 [-128.00 to 0.00] | 44.00 [-99.00 to 99.00] | -29.00 [-50.00 to 335.00] | 2.00 [0.00 to 204.00] | -5.00 [-188.00 to 126.00] | 94.00 [-54.00 to 386.00] | -1.50 [-47.00 to 344.00]
  CD8-CD40L, DAY 10: number analyzed (Participants) | 17 | 17 | 20 | 18 | 22 | 16 | 17
  CD8-CD40L, DAY 10 | 0.00 [0.00 to 1.00] | 0.00 [-50.00 to 1.00] | 0.00 [-50.00 to 48.00] | 0.00 [0.00 to 103.00] | 0.00 [0.00 to 109.00] | 24.00 [-5.00 to 94.50] | 0.00 [0.00 to 0.00]
  CD8-CD40L, DAY 21: number analyzed (Participants) | 14 | 17 | 19 | 19 | 17 | 15 | 16
  CD8-CD40L, DAY 21 | 0.00 [-48.00 to 0.00] | 0.00 [-1.00 to 0.00] | 0.00 [-18.00 to 60.00] | 0.00 [0.00 to 0.00] | 0.00 [-48.00 to 0.00] | 0.00 [-86.00 to 62.00] | 0.00 [-76.00 to 45.00]
  CD8-CD40L, DAY 42: number analyzed (Participants) | 10 | 17 | 11 | 15 | 17 | 15 | 14
  CD8-CD40L, DAY 42 | 0.00 [-48.00 to 47.00] | 0.00 [-49.00 to 0.00] | 0.00 [-7.00 to 46.00] | 0.00 [0.00 to 81.00] | 0.00 [0.00 to 0.00] | 0.00 [-81.00 to 135.00] | 0.00 [-101.00 to 48.00]
  CD8-IFN-γ, DAY 10: number analyzed (Participants) | 17 | 17 | 20 | 18 | 22 | 16 | 17
  CD8-IFN-γ, DAY 10 | 0.00 [-24.00 to 48.00] | -35.00 [-102.00 to 0.00] | 0.00 [-87.00 to 105.50] | 0.00 [-3.00 to 50.00] | 0.00 [-50.00 to 73.00] | 0.00 [-100.50 to 135.00] | 0.00 [-42.00 to 49.00]
  CD8-IFN-γ, DAY 21: number analyzed (Participants) | 14 | 17 | 19 | 19 | 17 | 15 | 16
  CD8-IFN-γ, DAY 21 | 0.00 [-63.00 to 76.00] | -6.00 [-96.00 to 0.00] | 0.00 [-159.00 to 54.00] | 0.00 [0.00 to 105.00] | 0.00 [-96.00 to 73.00] | 0.00 [-50.00 to 74.00] | 0.00 [-24.50 to 25.00]
  CD8-IFN-γ, DAY 42: number analyzed (Participants) | 10 | 17 | 11 | 15 | 17 | 15 | 14
  CD8-IFN-γ, DAY 42 | -0.50 [-48.00 to 0.00] | 0.00 [-96.00 to 0.00] | 49.00 [-134.00 to 86.00] | 14.00 [0.00 to 140.00] | -50.00 [-96.00 to 67.00] | 0.00 [-50.00 to 120.00] | 0.00 [-124.00 to 124.00]
  CD8-IL-2, DAY 10: number analyzed (Participants) | 17 | 17 | 20 | 18 | 22 | 16 | 17
  CD8-IL-2, DAY 10 | -1.00 [-103.00 to 59.00] | 0.00 [-38.00 to 47.00] | 2.50 [-123.00 to 66.50] | 0.00 [-98.00 to 100.00] | 0.00 [-50.00 to 118.00] | 0.00 [-80.00 to 160.50] | 0.00 [-21.00 to 96.00]
  CD8-IL-2, DAY 21: number analyzed (Participants) | 14 | 17 | 19 | 19 | 17 | 15 | 16
  CD8-IL-2, DAY 21 | -28.00 [-151.00 to 0.00] | 0.00 [-38.00 to 50.00] | -1.00 [-205.00 to 113.00] | 0.00 [0.00 to 129.00] | 0.00 [-81.00 to 38.00] | 0.00 [-60.00 to 98.00] | 0.00 [-16.00 to 78.50]
  CD8-IL-2, DAY 42: number analyzed (Participants) | 10 | 17 | 11 | 15 | 17 | 15 | 14
  CD8-IL-2, DAY 42 | -69.50 [-106.00 to 97.00] | 0.00 [-69.00 to 0.00] | 0.00 [-46.00 to 247.00] | 0.00 [-67.00 to 112.00] | 0.00 [-13.00 to 98.00] | 46.00 [-102.00 to 292.00] | 0.00 [-45.00 to 147.00]
  CD8-TNF-α, DAY 10: number analyzed (Participants) | 17 | 17 | 20 | 18 | 22 | 16 | 17
  CD8-TNF-α, DAY 10 | 4.00 [-99.00 to 99.00] | 0.00 [-97.00 to 47.00] | 23.00 [-49.50 to 121.00] | 0.00 [-48.00 to 194.00] | -3.00 [-140.00 to 46.00] | -24.50 [-127.50 to 114.50] | 0.00 [0.00 to 47.00]
  CD8-TNF-α, DAY 21: number analyzed (Participants) | 14 | 17 | 19 | 19 | 17 | 16 | 17
  CD8-TNF-α, DAY 21 | -10.50 [-97.00 to 21.00] | 0.00 [-50.00 to 75.00] | -7.00 [-127.00 to 114.00] | 0.00 [-45.00 to 247.00] | 0.00 [-49.00 to 47.00] | -24.50 [-127.50 to 114.50] | 0.00 [0.00 to 47.00]
  CD8-TNF-α, DAY 42: number analyzed (Participants) | 10 | 17 | 11 | 15 | 17 | 15 | 14
  CD8-TNF-α, DAY 42 | 0.00 [-99.00 to 47.00] | 48.00 [-69.00 to 159.00] | 74.00 [-7.00 to 289.00] | 0.00 [-52.00 to 255.00] | 0.00 [-62.00 to 149.00] | 99.00 [-34.00 to 243.00] | 24.00 [-95.00 to 120.00]

19. Primary Outcome: Serum HI Antibody Titers Against the Influenza A Virus Strain Subtype H9N2 (Anti-H9N2)
Description: Anti-H9N2 antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 21 post Dose 2 (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Titers | 55.9 [40.1 to 77.8] | 36.0 [25.8 to 50.2] | 31.0 [21.3 to 45.1] | 20.0 [15.2 to 26.2] | 63.1 [45.3 to 87.9] | 38.0 [26.7 to 54.1] | 26.0 [20.0 to 34.0]

20. Primary Outcome: Serum HI Antibody Titers Against the Influenza A Virus Strain Subtype H9N2 (Anti-H9N2)
Description: Anti-H9N2 antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 21 post Dose 3 (Day 210 for Subset 1 groups and Day 386 for Subset 2 groups)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 26 | 25 | 27 | 27 | 26 | 25 | 23 | 22 | 22 | 22 | 20 | 23 | 24 | 23
Titers | 49.5 [31.8 to 77.4] | 51.3 [30.4 to 86.7] | 51.1 [32.8 to 79.5] | 32.2 [21.8 to 47.5] | 71.0 [50.0 to 100.7] | 44.0 [30.3 to 64.0] | 28.3 [18.9 to 42.4] | 103.0 [63.3 to 167.5] | 41.3 [27.1 to 62.7] | 41.9 [23.7 to 74.1] | 21.4 [14.5 to 31.6] | 108.1 [69.4 to 168.5] | 62.5 [40.9 to 95.3] | 54.9 [37.4 to 80.5]

21. Primary Outcome: Number of Seroconverted Subjects Against Influenza A Subtype H9N2
Description: Seroconversion rate was defined as the percentage of vaccinees who had a pre-vaccination HI titer < 1:10 and a post-vaccination titre ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and a minimum four-fold increase in postvaccination titer
Time Frame: At Day 21 post Dose 2 (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Participants | 31 | 22 | 22 | 11 | 28 | 22 | 16

22. Primary Outcome: Number of Seroconverted Subjects Against Influenza A Subtype H9N2
Description: as for outcome 4
Time Frame: At Day 21 post Dose 3 (Day 210 for Subset 1 groups and Day 386 for Subset 2 groups)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 22 | 25 | 27 | 27 | 26 | 25 | 23 | 22 | 22 | 22 | 20 | 23 | 24 | 23
Participants | 15 | 18 | 19 | 13 | 20 | 15 | 10 | 19 | 10 | 12 | 4 | 17 | 15 | 14

23. Primary Outcome: Seroconversion Factor for Influenza A Subtype H9N2
Description: Seroconversion factor defined as the fold increase in serum HI GMTs on day 21 post Dose 3 (Day 42) compared to day 0.
Time Frame: At Day 21 post Dose 2 (Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Fold change | 6.3 [4.3 to 9.0] | 4.9 [3.5 to 6.8] | 4.3 [2.9 to 6.4] | 2.9 [2.3 to 3.7] | 8.3 [5.8 to 11.9] | 4.9 [3.4 to 7.2] | 3.7 [2.8 to 4.9]

24. Primary Outcome: Seroconversion Factor for Influenza A Subtype H9N2
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs on day 21 post Dose 3 (Day 210 for Subset 1 and Day 386 for Subset 2) compared to day 0.
Time Frame: At Day 21 post Dose 3 (Day 210 for Subset 1 groups and Day 386 for Subset 2 groups)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Fold change
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 26 | 25 | 27 | 27 | 26 | 25 | 23 | 22 | 22 | 22 | 20 | 23 | 24 | 23
Fold change | 5.4 [3.6 to 8.2] | 8.3 [5.1 to 13.5] | 7.9 [4.6 to 13.6] | 4.4 [3.1 to 6.4] | 10.5 [7.0 to 15.6] | 6.4 [4.3 to 9.6] | 4.3 [2.8 to 6.4] | 11.9 [6.4 to 21.9] | 5.5 [3.5 to 8.6] | 5.6 [3.2 to 9.6] | 2.8 [1.9 to 4.2] | 11.2 [5.9 to 21.1] | 2.0 [1.3 to 3.2] | 5.4 [3.0 to 9.9]

25. Primary Outcome: Number of Seroprotected Subjects Against H9N2
Description: as for outcome 7
Time Frame: At Day 21 post Dose 2 (Day 42)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group: | SB218352_8 Group: | SB218352_4 Group: | SB218352_2 Group: | SB218352_8AL Group: | SB218352_4AL Group: | SB218352_2AL Group:
Number analyzed (Participants) | 55 | 53 | 54 | 54 | 54 | 54 | 51
Participants | 41 | 27 | 27 | 14 | 35 | 25 | 19

26. Primary Outcome: Number of Seroprotected Subjects Against H9N2
Description: as for outcome 7
Time Frame: At Day 21 post Dose 3 (Day 210 for Subset 1 groups and Day 386 for Subset 2 groups)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 26 | 25 | 27 | 27 | 26 | 25 | 23 | 22 | 22 | 22 | 20 | 23 | 24 | 23
Participants | 18 | 18 | 21 | 17 | 22 | 18 | 11 | 20 | 13 | 13 | 6 | 20 | 17 | 16

27. Primary Outcome: Number of Subjects With Seroprotection Power Against H9N2
Description: as for outcome 9
Time Frame: At Day 21 post Dose 2 (Day 42)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 22 | 25 | 26 | 25 | 25 | 25 | 23 | 21 | 22 | 20 | 18 | 20 | 24 | 20
Participants | 13 | 12 | 14 | 9 | 13 | 12 | 4 | 17 | 12 | 7 | 1 | 14 | 9 | 10

28. Primary Outcome: Number of Subjects With Seroprotection Power Against H9N2
Description: as for outcome 9
Time Frame: At Day 21 post Dose 3 (Day 210 for Subset 1 groups and Day 386 for Subset 2 groups)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 21 | 24 | 26 | 25 | 25 | 25 | 23 | 21 | 21 | 20 | 18 | 20 | 23 | 21
Participants | 13 | 17 | 20 | 15 | 21 | 18 | 11 | 20 | 12 | 11 | 4 | 17 | 16 | 15

29. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness, swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = pain which prevents normal everyday activities. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm).
Time Frame: During the 4-days post Dose 1 (Days 0-3), post Dose 2 (Days 21-24) and across these doses
Population: The analysis was performed on the Total Vaccinated Cohort (TVc) included all vaccinated subjects (for whom diary card was available).
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group | SB218352_8 Group | SB218352_4 Group | SB218352_2 Group | SB218352_8AL Group | SB218352_4AL Group | SB218352_2AL Group
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55 | 55
Participants
  Any Pain, Dose 1 | 8 | 3 | 6 | 2 | 8 | 8 | 8
  Grade 3 Pain, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness (mm), Dose 1 | 7 | 4 | 3 | 1 | 10 | 6 | 5
  Grade 3 Redness (mm), Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling (mm), Dose 1 | 4 | 1 | 4 | 1 | 8 | 4 | 7
  Grade 3 Swelling (mm), Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2 | 7 | 4 | 4 | 2 | 5 | 4 | 6
  Grade 3 Pain, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness (mm), Dose 2 | 3 | 3 | 3 | 2 | 4 | 3 | 4
  Grade 3 Redness (mm), Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling (mm), Dose 2 | 2 | 1 | 3 | 2 | 3 | 4 | 2
  Grade 3 Swelling (mm), Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 12 | 7 | 9 | 4 | 10 | 9 | 9
  Grade 3 Pain, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness (mm), Across doses | 8 | 5 | 5 | 2 | 11 | 8 | 7
  Grade 3 Redness (mm), Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling (mm), Across doses | 5 | 2 | 6 | 2 | 10 | 5 | 7
  Grade 3 Swelling (mm), Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: as for outcome 29
Time Frame: During the 4 Days post Dose 3 (Days 189-192 for Subset 1 groups and Days 365-368 for Subset 2 groups)
Population: The analysis was performed on the Total Vaccinated Cohort (TVc) of Subsets, which included all vaccinated subjects (for whom the diary card was available).
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 26 | 23 | 23 | 24 | 23 | 22 | 23 | 26 | 24
Participants
  Any Pain | 6 | 1 | 5 | 3 | 9 | 8 | 6 | 4 | 1 | 0 | 0 | 1 | 1 | 2
  Grade 3 Pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness (mm) | 5 | 3 | 2 | 3 | 4 | 5 | 3 | 3 | 1 | 0 | 0 | 1 | 1 | 3
  Grade 3 Redness (mm) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling (mm) | 4 | 1 | 2 | 4 | 4 | 7 | 4 | 3 | 1 | 0 | 0 | 0 | 2 | 2
  Grade 3 Swelling (mm) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature higher than (≥) 37.5 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of any solicited general symptom regardless of intensity grade or relationship to the study vaccination. Grade 3 symptom = symptoms that prevented normal activity. Grade 3 fever = axillary temperature higher than (>) 39°C. Related symptom = symptom assessed by the investigator as being casually related to the study vaccination.
Time Frame: During the 4-days (Day 0-3) post Dose 1
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group | SB218352_8 Group | SB218352_4 Group | SB218352_2 Group | SB218352_8AL Group | SB218352_4AL Group | SB218352_2AL Group
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55 | 55
Participants
  Any Arthralgia | 3 | 2 | 4 | 3 | 2 | 3 | 6
  Grade 3 Arthralgia | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Arthralgia | 0 | 1 | 1 | 1 | 0 | 1 | 2
  Any Fatigue | 3 | 2 | 4 | 0 | 1 | 4 | 3
  Grade 3 Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fatigue | 0 | 1 | 2 | 0 | 0 | 0 | 1
  Any Temperature (Axillary) (°C) | 1 | 1 | 1 | 0 | 0 | 0 | 1
  Grade 3 Temperature (Axillary) (°C) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Temperature (Axillary) (°C) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any Headache | 4 | 5 | 6 | 2 | 8 | 4 | 6
  Grade 3 Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Headache | 1 | 0 | 0 | 1 | 1 | 0 | 2
  Any Myalgia | 3 | 3 | 3 | 2 | 4 | 1 | 5
  Grade 3 Myalgia | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Myalgia | 1 | 2 | 1 | 1 | 0 | 0 | 1
  Any Shivering | 2 | 2 | 4 | 1 | 3 | 3 | 1
  Grade 3 Shivering | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Shivering | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Any Sweating | 4 | 2 | 3 | 0 | 3 | 1 | 2
  Grade 3 Sweating | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating | 0 | 0 | 1 | 0 | 0 | 0 | 1

32. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 31
Time Frame: During the 4-days post Dose 2 (Days 21-24)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group | SB218352_8 Group | SB218352_4 Group | SB218352_2 Group | SB218352_8AL Group | SB218352_4AL Group | SB218352_2AL Group
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55 | 55
Participants
  Any Arthralgia | 3 | 2 | 0 | 2 | 3 | 5 | 2
  Grade 3 Arthralgia | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Arthralgia | 1 | 1 | 0 | 0 | 0 | 1 | 1
  Any Fatigue | 3 | 3 | 1 | 0 | 1 | 1 | 2
  Grade 3 Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fatigue | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Any Temperature (Axillary) (°C) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Temperature (Axillary) (°C) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Temperature (Axillary) (°C) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache | 4 | 2 | 6 | 4 | 4 | 3 | 3
  Grade 3 Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Headache | 1 | 1 | 1 | 0 | 1 | 1 | 2
  Any Myalgia | 2 | 3 | 2 | 1 | 3 | 4 | 1
  Grade 3 Myalgia | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Myalgia | 1 | 1 | 1 | 0 | 1 | 1 | 0
  Any Shivering | 1 | 1 | 2 | 0 | 1 | 2 | 1
  Grade 3 Shivering | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Shivering | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Any Sweating | 1 | 1 | 1 | 2 | 1 | 1 | 2
  Grade 3 Sweating | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating | 0 | 0 | 0 | 0 | 0 | 0 | 1

33. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 31
Time Frame: During the 4-Days (Day 0-3) across doses 1 and 2
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Group | SB218352_8 Group | SB218352_4 Group | SB218352_2 Group | SB218352_8AL Group | SB218352_4AL Group | SB218352_2AL Group
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55 | 55
Participants
  Any Arthralgia | 3 | 2 | 4 | 5 | 4 | 7 | 6
  Grade 3 Arthralgia | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Arthralgia | 1 | 1 | 1 | 1 | 0 | 2 | 3
  Any Fatigue | 5 | 4 | 5 | 0 | 1 | 5 | 4
  Grade 3 Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fatigue | 0 | 2 | 2 | 0 | 0 | 0 | 1
  Any Temperature (Axillary) (°C) | 1 | 2 | 1 | 0 | 0 | 0 | 1
  Grade 3 Temperature (Axillary) (°C) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Temperature (Axillary) (°C) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any Headache | 7 | 6 | 11 | 6 | 11 | 6 | 7
  Grade 3 Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Headache | 2 | 1 | 1 | 1 | 2 | 1 | 3
  Any Myalgia | 3 | 4 | 5 | 3 | 5 | 4 | 5
  Grade 3 Myalgia | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Myalgia | 2 | 2 | 2 | 1 | 1 | 1 | 1
  Any Shivering | 2 | 3 | 5 | 1 | 3 | 4 | 2
  Grade 3 Shivering | 2 | 3 | 5 | 1 | 3 | 0 | 0
  Related Shivering | 1 | 0 | 1 | 0 | 0 | 1 | 0
  Any Sweating | 5 | 3 | 4 | 2 | 4 | 2 | 3
  Grade 3 Sweating | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating | 0 | 0 | 1 | 0 | 1 | 0 | 1

34. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axilar temperature higher than (≥) 37.5 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of any solicited general symptom regardless of intensity grade or relationship to the study vaccination. Grade 3 symptom = symptoms that prevented normal activity. Grade 3 fever = fever higher than (>) 39°C. Related symptom = symptom assessed by the investigator as being casually related to the study vaccination.
Time Frame: During the 4 Days post Dose 3 (Days 189-192 for Subset 1 groups and Days 365-368 for Subset 2 groups)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 26 | 23 | 23 | 24 | 23 | 22 | 23 | 26 | 24
Participants
  Any Arthralgia | 2 | 1 | 1 | 0 | 0 | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Arthralgia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Arthralgia | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fatigue | 1 | 0 | 0 | 2 | 3 | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 0
  Grade 3 Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fatigue | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Any Temperature | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Temperature | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Temperature | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache | 3 | 0 | 4 | 2 | 2 | 3 | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 2
  Grade 3 Headache | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Headache | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Any Myalgia | 2 | 1 | 2 | 0 | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0
  Grade 3 Myalgia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Myalgia | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Any Shivering | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
  Grade 3 Shivering | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Shivering | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Any Sweating | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
  Grade 3 Sweating | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

35. Secondary Outcome: Number of Subjects With Unsolicited AEs
Description: as for outcome 11
Time Frame: During the 30-days post Dose 3 (Days 189-219 for Subset 1 groups and Days 365-395 for Subset 2 groups)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 26 | 23 | 23 | 24 | 23 | 22 | 23 | 26 | 24
Participants
  Any unsolicited AEs | 2 | 2 | 3 | 4 | 1 | 1 | 5 | 1 | 2 | 0 | 0 | 0 | 1 | 2
  Grade 3 unsolicited AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Related unsolicited AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 12
Time Frame: Within the 365-day post-vaccination period (Days 0-364 for Subset 1 groups) and within the 395-day post-vaccination period (Days 0-394 for Subset 2 groups)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 26 | 23 | 23 | 24 | 23 | 22 | 23 | 26 | 24
Participants
  Any SAEs | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Grade 3 SAEs: number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 26 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 SAEs | 1 | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  |  |  |  |
  Related SAEs: number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 26 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  |  |  |  |

37. Secondary Outcome: Number of Subjects With Any SAEs
Description: A SAE was any untoward medical occurrence which resulted in death, was life-threatening, resulted in hospitalization or prolongation of hospitalization, resulted in permanent of serious physical disability or incapacity, caused a congenital anomaly or birth defect in the offspring of a subject or might have put the subject at risk based on medical or scientific judgment or necessitated intervention to prevent such an event (e.q. invasive or malignant cancers, intensive treatment in an emergency room or at home for bronchospasm, blood dyscrasias, or convulsion that do not resulted in hospitalization). Only Subset 2 groups had available data for the specified time frame.
Time Frame: Up to 30-day post Dose 3 (Days 365-394)
Population: The analysis was performed on the Total Vaccinated Cohort (TVc) of Subset 2, which included all vaccinated subjects (for whom the diary card was available).
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 23 | 24 | 23 | 22 | 23 | 26 | 24
Participants | 0 | 2 | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Number of Subjects With Antibody Persistence
Description: Antibody persistence was evaluated in terms of seroprotection rate (SPR) against influenza A subtype H9N2 and seroconversion rate (SCR) against influenza A subtype H9N2.
Time Frame: At Days 189 and 365
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 26 | 25 | 23 | 22 | 23 | 22 | 20 | 23 | 25 | 23
Participants
  SPR, Day 189 | 13 | 9 | 11 | 6 | 8 | 10 | 3 | 12 | 7 | 5 | 2 | 14 | 7 | 5
  SPR, Day 365: number analyzed (Participants) | 27 | 26 | 27 | 27 | 26 | 25 | 23 | 22 | 22 | 22 | 20 | 23 | 24 | 23
  SPR, Day 365 | 13 | 14 | 10 | 7 | 11 | 6 | 4 | 20 | 13 | 13 | 6 | 20 | 17 | 16
  SCR, Day 189 | 8 | 9 | 9 | 4 | 6 | 7 | 3 | 10 | 6 | 5 | 0 | 9 | 5 | 2
  SCR, Day 365: number analyzed (Participants) | 27 | 26 | 27 | 27 | 26 | 25 | 23 | 22 | 22 | 22 | 20 | 23 | 24 | 23
  SCR, Day 365 | 8 | 13 | 8 | 5 | 10 | 5 | 2 | 19 | 10 | 12 | 4 | 17 | 15 | 14

39. Secondary Outcome: Seroconversion Factor (SCF) for Influenza A Subtype H9N2.
Description: SCF was defined as the fold increase in serum HI GMTs at the post-vaccination time points compared to Day 0, for each vaccine strain.
Time Frame: At Days 189 and 365
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | SB218352_15 Subset 1 | SB218352_8 Subset 1 | SB218352_4 Subset 1 | SB218352_2 Subset 1 | SB218352_8AL Subset 1 | SB218352_4AL Subset 1 | SB218352_2AL Subset 1 | SB218352_15 Subset 2 | SB218352_8 Subset 2 | SB218352_4 Subset 2 | SB218352_2 Subset 2 | SB218352_8AL Subset 2 | SB218352_4AL Subset 2 | SB218352_2AL Subset 2
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 26 | 25 | 23 | 22 | 23 | 22 | 20 | 23 | 25 | 23
fold increase
  SCF, Day 189 | 2.9 [1.9 to 4.5] | 3.4 [2.2 to 5.2] | 3.7 [2.1 to 6.5] | 2.3 [1.7 to 3.1] | 3.2 [2.1 to 5.0] | 3.2 [2.1 to 4.9] | 1.8 [1.3 to 2.5] | 3.3 [1.8 to 6.1] | 2.7 [1.5 to 4.9] | 2.1 [1.1 to 4.1] | 1.5 [1.1 to 1.9] | 5.8 [3.4 to 10.0] | 2.2 [1.3 to 3.8] | 1.7 [1.1 to 2.8]
  SCF, Day 365: number analyzed (Participants) | 27 | 26 | 27 | 26 | 26 | 25 | 23 | 22 | 22 | 22 | 20 | 23 | 24 | 23
  SCF, Day 365 | 3.1 [2.1 to 4.6] | 5.4 [3.5 to 8.5] | 4.3 [2.5 to 7.4] | 2.1 [1.4 to 3.0] | 4.3 [3.0 to 6.1] | 2.9 [1.9 to 4.2] | 2.1 [1.4 to 3.1] | 11.9 [6.4 to 21.9] | 5.5 [3.5 to 8.6] | 5.6 [3.2 to 9.6] | 2.8 [1.9 to 4.2] | 11.2 [5.9 to 21.1] | 7.5 [4.9 to 11.5] | 5.4 [3.0 to 9.9]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: up to Day 51.
Description: One subject from the SB218352_15 Group reported both SAE(s) included in the Adverse Events section.
Arm/Group | SB218352_15 Group | SB218352_8 Group | SB218352_4 Group | SB218352_2 Group | SB218352_8AL Group | SB218352_4AL Group | SB218352_2AL Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/55 | 0/55 | 0/55 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/55 | 0/55 | 1/55 | 0/55 | 0/55 | 0/55 | 1/55
Other Adverse Events (participants affected / at risk) | 26/55 | 16/55 | 25/55 | 14/55 | 28/55 | 22/55 | 24/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB218352_15 Group (N=55) | SB218352_8 Group (N=55) | SB218352_4 Group (N=55) | SB218352_2 Group (N=55) | SB218352_8AL Group (N=55) | SB218352_4AL Group (N=55) | SB218352_2AL Group (N=55)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB218352_15 Group (N=55) | SB218352_8 Group (N=55) | SB218352_4 Group (N=55) | SB218352_2 Group (N=55) | SB218352_8AL Group (N=55) | SB218352_4AL Group (N=55) | SB218352_2AL Group (N=55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (5) | 5 (5) | 5 (5) | 4 (5) | 8 (11) | 6 (9)
Chills (General disorders) | 2 (3) | 4 (4) | 5 (8) | 1 (1) | 4 (5) | 5 (6) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 9 (15) | 7 (10) | 6 (8) | 3 (6) | 13 (18) | 9 (14) | 7 (12)
Fatigue (General disorders) | 5 (7) | 4 (5) | 5 (5) | 2 (2) | 4 (5) | 6 (7) | 6 (7)
Headache (Nervous system disorders) | 8 (11) | 6 (7) | 13 (16) | 8 (8) | 12 (14) | 7 (10) | 8 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 4 (5) | 2 (2) | 5 (5) | 2 (2) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 5 (7) | 5 (7) | 3 (3) | 6 (8) | 6 (8) | 5 (6)
Pain (General disorders) | 16 (21) | 8 (8) | 13 (15) | 6 (7) | 14 (22) | 14 (20) | 12 (20)
Swelling (General disorders) | 7 (10) | 3 (3) | 6 (9) | 4 (7) | 13 (15) | 10 (15) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.